CLINICAL TRIAL: NCT02241564
Title: Follow-up of Malignancies in Transplanted Patients
Brief Title: Malignancies in Transplanted Patients
Acronym: MALTX
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Tomas Lorant, Associate professor, Uppsala University
Other Study IDs: MALTX-001
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
Keywords: Immunosuppression
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Malignancy post transplantation
  Interventions: Other: Referral to a multidisciplinary expert panel at the Uppsala University Hospital after tumor detection; Drug: Switch from calcineurin inhibitor to an mTOR inhibitor

INTERVENTIONS:
Other: Referral to a multidisciplinary expert panel at the Uppsala University Hospital after tumor detection
Drug: Switch from calcineurin inhibitor to an mTOR inhibitor

SUMMARY:
The aim of the project is to improve the overall treatment and outcome of renal, pancreas or liver transplanted patients who have encountered a malignancy by a structured treatment program for diagnosis and treatment of the malignancy, optimization of the immunosuppressive treatment, follow-up and evaluation of the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and capable of giving written informed consent of participation in the project
* Patients with a previous diagnosed or presently diagnosed or reoccurrence of a malignancy (other then basal cell carcinoma)

Exclusion Criteria:

* Patients with a primary liver cancer as cause of the transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney, pancreas or liver transplanted patients in the Uppsala/Örebro region with a diagnosed malignancy pre or post transplantation
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2007-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Patient survival | 12 months, 2 years, 3 years
  After inclusion

SECONDARY OUTCOMES:
Graft survival | 12 months, 2 years, 3 years
  After inclusion
ImmuKnow Assay value | 12 months
Tumour progression/regression/reoccurrence | 12 months, 2 years, 3 years
Maintained switch of immunosuppression from calcineurin inhibitor to mTOR inhibitor | 3 years
Kidney function | 12 months, 2 years, 3 years
  Creatinine measure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Section of Transplantation Surgery, Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Hellstrom V, Lorant T, Dohler B, Tufveson G, Enblad G. High Posttransplant Cancer Incidence in Renal Transplanted Patients With Pretransplant Cancer. Transplantation. 2017 Jun;101(6):1295-1302. doi: 10.1097/TP.0000000000001225. PMID 27163539
- [Derived] Hellstrom VC, Enstrom Y, von Zur-Muhlen B, Hagberg H, Laurell A, Nyberg F, Backman L, Opelz G, Dohler B, Holmberg L, Tufveson G, Enblad G, Lorant T. Malignancies in transplanted patients: Multidisciplinary evaluation and switch to mTOR inhibitors after kidney transplantation - experiences from a prospective, clinical, observational study. Acta Oncol. 2016 Jun;55(6):774-81. doi: 10.3109/0284186X.2015.1130855. Epub 2016 Jan 29. PMID 26824275